CLINICAL TRIAL: NCT04023253
Title: Comparisons of the Impact of Beta-3 Agonist Versus Antimuscarinics on Psychological Distress, Sexual Function, Bladder Wall Thickness and Blood Flow in Women With Overactive Bladder Syndrome: a Randomized Controlled Study.
Brief Title: Pharmacologic Effect for Female Overactive Bladder Syndrome: Mirabegron Versus Solifenacin
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Responsible Party: Principal Investigator, Sheng-Mou Hsiao, Chief and Associate Professor, Department of Obstetrics and Gynecology, Far Eastern Memorial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 108003-F
Record Dates: First submitted 2019-07-12; First posted 2019-07-17 (Actual); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Overactive Bladder Syndrome
MeSH Terms: interventions — mirabegron; Solifenacin Succinate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- mirabegron (Experimental): Receive mirabegron 2 mg treatment per day
  Interventions: Drug: Mirabegron
- solifenacin (Experimental): Receive solifenacin 5 mg treatment per day
  Interventions: Drug: Solifenacin

INTERVENTIONS:
Drug: Mirabegron — Mirabegron 25 mg
  Arms: mirabegron
Drug: Solifenacin — Solifenacin 5 mg
  Arms: solifenacin

SUMMARY:
To assess the impact of mirabegron versus solifenacin on psychological distress, sexual function, bladder wall thickness and bladder blood flow.

DETAILED DESCRIPTION:
To assess the impact of mirabegron versus solifenacin on psychological distress, sexual function, bladder wall thickness and blood flow.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder syndrome

Exclusion Criteria:

* Allergy to mirabegron or solifenacin.
* Patients with severe hypertension who are difficult to control, known urethral diverticulum, known bladder malignant tumors, urinary retention patients, gastric retention patients, uncontrolled angular glaucoma patients, dialysis patients, severe renal dysfunction , moderate liver dysfunction, use strong inhibitors of CYP3A4 such as ketoconazole.

Min Age: 20 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Global response assessment | 12 weeks
  Between-group difference in the score of Global response assessment

SECONDARY OUTCOMES:
Total score of Brief Symptoms Rating Scales | 12 weeks
  Between-group difference in the changes of total score of Brief Symptoms Rating Scales
Female sexual function index | 12 weeks
  Between-group difference in the changes of total score of female sexual function index
Bladder wall thickness | 12 weeks
  Between-group difference in the changes of bladder wall thickness
Blood flow index of the bladder | 12 weeks
  Between-group difference in the changes of blood flow index of the bladder

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Obstetrics and Gynecology, Far-Eastern Memorial Hospital, Banqiao District, New Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No